CLINICAL TRIAL: NCT04951908
Title: Correlation Between Types of Lateral Pterygoid Muscle Attachment, Type of Disk Displacement and Osteoarthritic Changes of the Temporomandibular Joint
Brief Title: Correlation Between Types of Lateral Pterygoid Muscle Attachment and Internal Derangement of the Temporomandibular Joint
Acronym: LPM & TMJ
Status: Completed | Type: Observational
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ayman Hegab, associate professor of oral and maxillofacial surgery, Al-Azhar University
Other Study IDs: AUAREC20190511-11
Record Dates: First submitted 2021-06-29; First posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-06

CONDITIONS: TMJ Disorder
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control group: NORMAL TMJ
  Interventions: Diagnostic Test: MRI
- Study group: Patients with TMJ internal derangement
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — MRI of TMJ

SUMMARY:
the study aimed to evaluate the clinical and MRI finding of TMJ AND LPM with predication of the risk factors. Study design: this retrospective study included 1365 joints in 800 patients diagnosed as TMJ internal derangement and all the patients examined by MRI from 2008 to 2019. Cases with loss of continuity of articular disk or the posterior attachment of the disk were considered as positive cases.

DETAILED DESCRIPTION:
the study aimed to evaluate the clinical and MRI finding of TMJ with LPM with predication of the risk factors. Study design: this retrospective study included patients diagnosed as TMJ internal derangement and all the patients examined by MRI from 2008 to 2019. Cases with loss of continuity of articular disk or the posterior attachment of the disk were considered as positive cases.

ELIGIBILITY:
Inclusion Criteria:

- study included patients seeking treatment for TMD at Al-Azhar University Hospital and the outpatient clinic at the Faculty of Dental Medicine of Al-Azahr University.

Exclusion Criteria:

* Exclusion Inclusion criteria: Patients were included if they were older than 18 years and diagnosed with TMJD. criteria for this study included systemic diseases (the presence of polyarthritis or other rheumatic diseases), contraindications for MRI (e.g., implanted metal or medical devices, claustrophobia), the presence of neurologic disorders, head and neck cancer, oral submucous ﬁbrosis, a history of TMJ surgery, a history of previous nonsurgical treatment such as occlusal splints, and a history of joint injection with HA/PRP. Trauma patients with subcondylar fracture and patients with congenital and developmental disorders of the TMJ were also excluded from the study.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The retrospective study included patients seeking treatment for TMD at Al-Azhar University Hospital and the outpatient clinic at the Faculty of Dental Medicine of Al-Azahr University. The sample originally included patients who provided consent to participate in this study and who ultimately underwent treatment for TMJD between 2008 and 2019.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Actual)
Dates: Start 2019-11-30 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
VAS | baseline (pre treatment)
  pain index scores were measured using a 10-point visual analogue scale (VAS), with 0 indicating absence of pain and 10 indicating the worst pain.
mouth opening | baseline (pre treatment)
  maximum nonassisted (voluntary) mouth opening (MVMO) in millimetres

SECONDARY OUTCOMES:
joint sound | baseline (pre treatment)
  and the joint sound was then determined by combining 3 means: (1) palpation of the TMJ zone by the clinician, (2) the patient's self-reporting regarding whether the joint sound could be heard, and (3) auscultation of the TMJ zone with the stethoscope.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dental Medicine Alazhar University, Cairo, Nasr City, Egypt

IPD SHARING:
Plan to Share IPD: No